CLINICAL TRIAL: NCT05645133
Title: Evaluation of a Pediatric Reference Interval Using QPLUS System
Brief Title: QPlus Pediatric Reference Interval
Status: Terminated | Type: Observational
Why Stopped: PI relocated to another institution
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IIS-005
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Pediatric ALL; Healthy
Keywords: QPlus; Quantra; Pediatric; Reference Range
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Diagnostic Test — Diagnostic device to monitor coagulation properties of a whole blood sample at the point of care
  Other Names: Point of Care test; Quantra

SUMMARY:
Evaluation of coagulation results reported by the Qplus Quantra System to determine pediatric reference range intervals.

DETAILED DESCRIPTION:
Single center observational study of the pediatric patient population (< 18yrs) with normal coagulation function to determine the reference range interval for the clotting parameters reported by the Quantra QPlus system.

ELIGIBILITY:
Inclusion Criteria:

* <18yrs
* Scheduled for procedure requiring anesthesia
* Access to blood sampling
* Consented

Exclusion Criteria:

* >18yrs of age
* pre-term babies
* patients with know hematological disorders
* Difficult to obtain blood sampling
* Has received a blood product transfusion within the last 24hrs.
* Legal guardian unwilling to consent

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients with normal coagulation function who have been scheduled to undergo a procedure and blood sampling access has been established. All genders, racial and ethnic profiles will be described.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Reference range interval for measurement of clot time (CT) parameter | Baseline, after access placement before any procedures
  Reference range interval determined in this study will serve as the reference for CT results in this particular population
Reference range interval for measurement of clot time (CTH) parameter | Baseline, after access placement before any procedures
  Reference range interval determined in this study will serve as the reference for CTH results in this particular population
Reference range interval for measurement of clot stiffness (CS) parameter | Baseline, after access placement before any procedures
  Reference range interval determined in this study will serve as the reference for CS results in this particular population
Reference range interval for measurement of Fibrinogen Contribution to clot stiffness (FCS) parameter | Baseline, after access placement before any procedures
  Reference range interval determined in this study will serve as the reference for FCS results in this particular population
Reference range interval for measurement of Platelet Contribution to clot stiffness (PCS) parameter | Baseline, after access placement before any procedures
  Reference range interval determined in this study will serve as the reference for PCS results in this particular population

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Tirotta, MD, Principal Investigator — Nicklaus Childrens
Locations (1):
- Nicklaus Childrens Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No